CLINICAL TRIAL: NCT00496652
Title: DAHANCA 19: A Randomized Study of the Importance of the EGFr-Inhibitor Zalutumumab for the Outcome After Primary Curative Radiotherapy for Squamous Cell Carcinoma of the Head and Neck
Brief Title: DAHANCA 19: The Importance of the EGFr-inhibitor Zalutumumab for the Outcome After Curative Radiotherapy for HNSCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Danish Head and Neck Cancer Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAHANCA 19; Ethical Comittee: 20070091; DKMA: 2612-3486
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Cancer of the Head and Neck
Keywords: Squamous Cell Carcinomas of the Head and Neck; Epidermal Growth Factor receptor; Antibody; Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy; zalutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Radiotherapy (+cisplatin to stage 3+4)
  Interventions: Radiation: Radiotherapy
- 2 (Experimental): Radiotherapy 66-68 Gy, 2Gy/fx, 6 fx/week (+ weekly cisplatin 40 mg/m2 during radiotherapy to stage 3+4) + Zalutumumab 8 mg/kg every week during radiotherapy + the week before start of radiotherapy (as loading dose)
  Interventions: Drug: Zalutumumab

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy 66-68 Gy, 2Gy/fx, 6 fx/week (+ weekly cisplatin 40 mg/m2 during radiotherapy to stage 3+4)
  Arms: 1
Drug: Zalutumumab — Zalutumumab 8 mg/kg every week during radiotherapy + the week before start of radiotherapy (as loading dose)
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the addition of the fully human EGFr antibody zalutumumab to primary curative radiotherapy increases locoregional control in Squamous Cell Carcinomas of the Head and Neck.

DETAILED DESCRIPTION:
Radiotherapy to Squamous Cell Carcinomas of the Head and Neck have been modified during the last decades by altered fractionation, the addition of concomitant chemotherapy or modification of hypoxia. By these modifications the locoregional control, disease-specific survival or overall survival have been increased but the price have been increased morbidity.

The addition of antibodies against the Epidermal Growth Factor receptor (EGFR-I) may further increase the control and survival of patients with Squamous Cell Carcinomas of the Head and Neck when combined with radiotherapy and/or chemotherapy.

The aim of the present study is to determine whether

1. The addition af the EGFr-I zalutumumab increases locoregional control in Squamous Cell Carcinomas of the Head and Neck
2. Whether disease-specific survival or overall survival is improved by addition of zalutumumab
3. Whether the addition of zalutumumab to primary curative radiotherapy or chemoradiotherapy is feasible and tolerable
4. Acute and late toxicity to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven squamous cell carcinoma of the pharynx, larynx (excp. stage 1 larynx and stage 1+2 glottic larynx)
* Curative intent and no prior treatment
* Age > 18 years
* WHO performance 0-2 (incl.)
* No prior treatment with EGFr-I
* Informed consent according to local guidelines and national law
* The patient is able (psychological, sociological, geographical and physical) to carry through the treatment and follow-up
* Fertile women must use contraceptive devices (IUD or oral contraceptives)

Exclusion Criteria:

* Rhinopharynx or carcinomas of unknown origin
* Distal metastases
* Other malignant diseases (prior or current) except from planocellular skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2007-11; Primary Completion 2012-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Locoregional control after curative intended radiotherapy/chemoradiotherapy +/- zalutumumab | 5 years

SECONDARY OUTCOMES:
Disease-specific survival and overall control Acute and late toxicity | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jens Overgaard, Prof. MD, Principal Investigator — Danish Head and Neck Cancer Group (DAHANCA)
Locations (1):
- Department of Experimental Clinical Oncology, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- See also: official webpage of the Danish Head and Neck Cancer Group (DAHANCA) — http://www.dahanca.dk